CLINICAL TRIAL: NCT00005348
Title: Adipose Distribution and Atherosclerosis
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 4217; R01HL046208 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-04

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Carotid Stenosis
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Carotid Stenosis

SUMMARY:
To relate distribution of adipose tissue measured by a then new imaging technique, Magnetic Resonance Imaging (MRI) to extracranial carotid atherosclerosis, cardiovascular disease risk factors, and to more conventional measures of fat distribution such as body mass index (BMI) and waist/hip ratio. The primary hypothesis was that patients with extracranial carotid atherosclerosis (cases) had more intra-abdominal fat and a higher ratio of intra-abdominal fat to total or subcutaneous fat than age-sex-race matched controls.

DETAILED DESCRIPTION:
BACKGROUND:

The study was ancillary to an NIH funded population-based project, the Atherosclerosis Risk in Communities Study (ARIC) that is ongoing in Forsyth County, North Carolina.

DESIGN NARRATIVE:

Using MRI, the investigators sought to demonstrate strong relationships between intra-abdominal fat and a number of cardiovascular disease risk factors, including history of hypertension, diabetes, cigarette smoking, family history of cardiovascular disease, plasma concentrations of triglyceride, high density lipoprotein (HDL) cholesterol, HDL2 cholesterol, apo A1, Apo B, postprandial lipid response to a fat rich meal, glucose, insulin, sex hormone binding globulin, and total and free testosterone. Certain other risk factors were less certain to show a relation to intra-abdominal fat as measured by MRI, including various hemostatic factors, as well as certain dietary factors such as consumption of alcohol, dietary fat, and cholesterol, but this research afforded an opportunity to explore these relationships. Finally, the investigators proposed to relate intra-abdominal fat to more conventional measures of fat distribution (waist/hip ratio, subscapular skinfold thickness, etc.) in an attempt to identify strong correlates of intra-abdominal fat that could be more easily measured.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) recor

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1991-04; Study Completion 1993-03 (Actual)

REFERENCES:
- [Background] Terry JG, Hinson WH, Evans GW, Schreiner PJ, Hagaman AP, Crouse JR 3rd. Evaluation of magnetic resonance imaging for quantification of intraabdominal fat in human beings by spin-echo and inversion-recovery protocols. Am J Clin Nutr. 1995 Aug;62(2):297-301. doi: 10.1093/ajcn/62.2.297. PMID 7625335